CLINICAL TRIAL: NCT03479034
Title: A Prospective Qualitative and Quantitative Controlled Study, Exploring the Impact of Patient Centred Digital Prescriptions on Health, in Patients With Chronic Health Conditions
Brief Title: Patients Empowered With Digital Scripts: ScalaMed
Acronym: PEDS
Status: Withdrawn | Type: Observational
Why Stopped: Investigator decided not to proceed in Australia at this stage.
Sponsor: Holdsworth House Medical Practice (Other)
Collaborators: ScalaMed (Unknown)
Responsible Party: Sponsor
Other Study IDs: SCALA001
Record Dates: First submitted 2018-01-21; First posted 2018-03-27 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Technology
Keywords: digital; prescription; Application

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: * Ages 18-85
  * Cognitively able to understand instructions and care for themselves
  * Lives in the community (not institutionalised)
  * Owner of a smartphone and able to use Apps
  * On 3 or more chronic prescription medications
  * Has had experience with prescriptions in Australia for at least 1 year
  * Current patient attending Holdsworth House Medical Practice
  Willing to use the ScalaMed ePrescription application
  Interventions: Other: ScalaMed ePrescription application

INTERVENTIONS:
Other: ScalaMed ePrescription application — Mobile phone application (Android and Apple) for storing electronic prescriptions

SUMMARY:
A prospective qualitative and quantitative controlled study, exploring the impact of patient centred digital prescriptions on health, in patients with chronic health conditions.

DETAILED DESCRIPTION:
ScalaMed is an innovative new consumer centred solution for securing prescriptions through a blockchain solution - a cryptographic distributed database, that can give consumer access to their prescriptions at all times. It aims to solve interoperability challenges that exist in healthcare, by creating a ledger of prescriptions, and giving consumers access to this information to own and share as they need. The solution will be accessed through an application available on a smart phone, will be fully compliant with security and privacy laws, and will be made available to consumers, clinicians, and pharmacies enrolled in this study free of charge. The system also allows patients to monitor the usage of their prescriptions - eg when they need a new one, and allows them to choose how and where they want to use their prescriptions like with paper.

This study will explore whether empowering consumers with their digital prescriptions in a digital format through a blockchain based methodology of storing and accessing their data, will improve the flow of clinically important information, improve the frequency of data sharing, improve the self-management of the patient, improve adherence to treatments, reduce interactions and adverse events associated with medications, reduce the burden on clinical practice, improve efficiency, reduce the amount of paper, increase consumer engagement and improve patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-85
* Cognitively able to understand instructions and care for themselves
* Lives in the community (not institutionalised)
* Owner of a smartphone and able to use Apps
* On 3 or more chronic prescription medications
* Informed consent as documented by signature (Appendix Informed Consent Form)
* Has had experience with prescriptions in Australia for at least 1 year
* For the clinicians - any clinician who is using the ScalaMed prescription system in the Holdsworth House
* For pharmacists - who are utilising the ScalaMed system in one of the four clinics

Exclusion Criteria:

* Known or suspected non-compliance, drug or alcohol abuse
* Inability to follow the procedures of the study due to language problems, psychological disorders, dementia of the participant
* Previous enrolment into the current study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients of Holdsworth House Medical Practice
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-01 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Patient preference | 6 months
  Primary outcome is the change from baseline in patient preference for ScalaMed over previous prescription management tools after 3-months, determined through a questionnaire using a 4 point Likert scale.
  9) I prefer Scalamed to my previous system of managing prescriptions
  1. Strongly agree
  2. Somewhat agree
  3. somewhat disagree
  4. strongly disagree

SECONDARY OUTCOMES:
Clinician prefence | 3 months
  The change from baseline in clinician preference for ScalaMed over previous prescription management tools after 3-months, determined through a questionnaire using a 4 point Likert scale.
  1. I prefer ScalaMed over paper for helping patients manage their prescriptions
  1. Strongly agree
  2. Somewhat agree
  3. somewhat disagree
  4. strongly disagree
Prescriber satisfaction | 6 months
  Outcome will be determined through a questionnaire and will describe prescriber satisfaction in managing patient's prescriptions at 6 months 19 questions in relation to the impact of electronic prescriptions on the patient's journey, from when a prescription is required to when their medicines are received with the options: Strongly Disagree, Slightly Disagree, Slightly Agree, Strongly Agree. For example:
  1. Easier for me to send patients prescriptions when they are not in the clinic
  2. Patients have increased control and understanding of their medicines
  3. Electronic prescriptions are more patient centric
Clinical Implications | 6 months
  Determined through a questionnaire, a description of the clinical implications associated with consumers utilizing digital prescriptions at 6 months Please indicate the extent to which you agree with the following statements about the impact of ScalaMed electronic prescriptions on patient care: Strongly Disagree, Slightly Disagree, Slightly Agree, Strongly Agree
  1. Reduces the likelihood of prescription errors
  2. Makes it easier for patients to have their prescriptions dispensed
  3. Empowers patients with their data
  4. Reduces admin burden in the clinic
  5. Reduces fraud
  6. Helps patients adhere to their medicine
  7. Integrates data across providers
  8. Reduces workload
  9. Reduced lost of missing prescriptions
Patient measures | 6 months
  Description of clinically relevant patient measures affected by proper utilization of medication information, measured through repeat questionnaires over 6 months
  1. Which of the following features of ScalaMed do you value? (Tick all that apply)
  1. No paper
  2. Value for patient - ease and convenience and source of truth data
  3. Ability to view patient's prescribing across doctors
  4. Ability to view patient's dispensing history
  5. Potential for interaction and allergy alerts
  6. Ability to send prescriptions to patients remotely (prescriber) / patients can send me prescriptions remotely (pharmacy)
Digital sharing | 6 months
  To describe the relationship of digitally sharing data and communications between the consumer and their care team, measured through repeat questionnaires over 6 months
Care implications | 6 months
  A description of the relationship between shared data and efficient and relevant care measured through a Combination of patient and clinical questionnaires over 6 months.
  Patients questionnaires:
  1. Did you find a mistake, or issue with a prescription that you were sent BECAUSE of ScalaMed - that is, ScalaMed helped you see that you received an incorrect medicine or dosage? Yes/No
  2. Did you see another health care practitioner since you last completed a questionnaire? Yes /No Did you show them your prescription data on ScalaMed? Yes/No Clinician Questions
  1.Which of the following features of ScalaMed do you value? (Tick all that apply) 2.Electronic prescriptions have the potential to reduce miscommunication between health professionals: Strongly Disagree, Slightly Disagree, Slightly Agree, Strongly Agree
Pharmacy engagement | 6 months
  A description of consumer engagement and experience at the pharmacy over 6 months, as measured by repeat questionnaires.
  Pharmacyexamples: 4 questions in relation to the impact of electronic prescriptions on the patient's journey, from when a prescription is required to when their medicines are received with the options: Strongly Disagree, Slightly Disagree, Slightly Agree, Strongly Agree. For example:
  d. Electronic prescriptions are more legible e. Has potential to reduce miscommunication between health professionals Patient examples:Since you last completed a questionnaire have you arrived in a pharmacy to find you had no more prescriptions/repeats available? Yes/no At the moment do you know where all your prescriptions are stored/kept? Yes/no

CONTACTS AND LOCATIONS:
Overall Officials: Tal Rapke, Dr, Study Director — ScalaMed

IPD SHARING:
Plan to Share IPD: No